CLINICAL TRIAL: NCT01335646
Title: Surgery Versus Standardized Non-operative Care for the Treatment of Lumbar Disc Herniations: A Canadian Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The London Spine Centre (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UWO16000
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Lumbar Spine Disc Herniation; Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Physical Therapy Modalities; Injections, Epidural; Educational Status; Anti-Inflammatory Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Surgery (Active Comparator)
  Interventions: Procedure: Lumbar Microdiscectomy
- Non-operative (Active Comparator)
  Interventions: Other: Physiotherapy, Epidural injections, Education, Pain Medications, Anti-inflammatories

INTERVENTIONS:
Procedure: Lumbar Microdiscectomy — lumbar discectomy within 1 month of randomization
  Arms: Surgery
Other: Physiotherapy, Epidural injections, Education, Pain Medications, Anti-inflammatories — Physiotherapy following standardized protocol Epidurals - Depomedrol 80 mg plus 10cc of 0.35% Lidocaine Education to occur at each visit Medications may include: NSAIDS; Acetaminophen with codeine or oxycodone or tramadol; Amitriptyline or Neurontin or Pregabalin
  Arms: Non-operative

SUMMARY:
The objective of this study is to determine if surgery is superior to non-operative care for sciatica caused by a lumbar disc herniation. This study will include patients that have had severe sciatica for greater than 4 months which reflects the wait time of the Canadian health care system. This study is an opportunity to make an important contribution to medical science as there is no "top tier" evidence for or against this highly prevalent surgery. Although there have been several recent randomized trials in the field, all have been marred by a large number of patient crossing over from non-operative to operative treatment. Due to the wait for spine surgery, the Canadian system has a built-in delay that prevents such a cross over of patients. This study capitalizes on this unique opportunity to perform a high caliber surgical trial. Patients consenting to be in the study will be randomly assigned to expedited surgery within three weeks or standardized non-operative care while they wait on the surgeons list for consultation and then surgery (minimum wait of 9 months). The study will assess pain, function, quality of life, satisfaction, and work status to determine if one treatment is superior.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 60 years old
2. Unilateral, single L5 or S1 radiculopathy (leg pain following dermatomal distribution of L5 or S1)

   * Leg dominant pain over central back pain
   * Positive straight leg raise <70 degrees
3. MRI with corresponding L4-5 or L5-S1 posterolateral disc herniation*
4. Radicular symptom duration greater than 4 months and less than 12 months. May be recurrent if first episode occurred within 12 months and duration of presenting episode is greater than 4 months.
5. Agree to possible discectomy

Exclusion Criteria:

1. Radiculopathy secondary to foraminal stenosis
2. Radiculopathy secondary to intra-foraminal or far lateral disc herniation
3. Radiculopathy secondary to lumbar central or lateral recess stenosis not caused by a posterolateral disc herniation
4. Previous lumbar surgery at involved level
5. Lumbar spondylolisthesis or lateral listhesis at level of disc herniation
6. Lumbar Scoliosis greater than 10 degrees

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2010-03-21 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for leg pain intensity | 6 months
  (Scale 0-10: 0 = no pain, 10 worst pain)

SECONDARY OUTCOMES:
Visual Analogue Scale for leg pain intensity | enrollment, 6 weeks, 3 months, 6 months, 1 year
  (Scale 0-10: 0 = no pain, 10 worst pain)
Visual Analogue Scale for central back pain intensity | enrollment, 6 weeks, 3 months, 6 months, 1 year
  (Scale 0-10: 0 = no pain, 10 worst pain)
Visual Analogue Scale for leg pain frequency | enrollment, 6 weeks, 3 months, 6 months, 1 year
  (Scale 0-10: 0 = no pain, 10 worst pain)
Visual Analogue Scale for central back pain frequency | enrollment, 6 weeks, 3 months, 6 months, 1 year
  (Scale 0-10: 0 = no pain, 10 worst pain)
Oswestry Disability Index | enrollment, 6 weeks, 3 months, 6 months, 1 year
  Scale 0-100; 0= no disability, 100 worst disability)
SF36 - Generic Health Outcome Measure | enrollment, 6 weeks, 3 months, 6 months, 1 year
  physical component summary score and mental component summary score, higher scores indicate better quality of life
Return to Work Status (% of patients employed) | enrollment, 6 weeks, 3 months, 6 months, 1 year
  Employed vs unemployed
Satisfaction with treatment (% of patients satisfied with treatment) | 6 weeks, 3 months, 6 months, 1 year
  satisfied vs unsatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Science Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Bailey CS, Rasoulinejad P, Taylor D, Sequeira K, Miller T, Watson J, Rosedale R, Bailey SI, Gurr KR, Siddiqi F, Glennie A, Urquhart JC. Surgery versus Conservative Care for Persistent Sciatica Lasting 4 to 12 Months. N Engl J Med. 2020 Mar 19;382(12):1093-1102. doi: 10.1056/NEJMoa1912658. PMID 32187469